CLINICAL TRIAL: NCT06816069
Title: Early Stage Safety and Efficacy Assessment for the Temporary Facial(both Cheeks) Skin Tightening Improvement Effect Using the Monopolar Radiofrequency Device: Prospective, Open-label, Single Center, Single-arm, Pilot Clinical Trial
Brief Title: Study on Safety and Efficacy of Monopolar Radio Frequency Device for Facial Skin Tightening
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CLASSYS Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VM-01
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Skin Aging
Keywords: VOLNEWMER; Monopolar radiofrequency device; MRF; Skin Tightening; Facial skin treatment; Skin Elasticity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- VOLNEWMER (Experimental): Each subject will undergo a procedure using VOLNEWMER's F-Tip or V-tip electrode with either the Basic mode or Easy mode, depending on the treatment area.
  Interventions: Device: VOLNEWMER

INTERVENTIONS:
Device: VOLNEWMER — Monopolar radiofrequency device

SUMMARY:
Objective:

The goal of this clinical trial is to evaluate the safety and efficacy of the VOLNEWMER monopolar radiofrequency device developed by CLASSYS Inc. This study is a prospective, single-center, single-arm, pilot clinical trial.

Research Questions:

1. Does the VOLNEWMER device improve skin elasticity?
2. Is the safety profile of the VOLNEWMER device acceptable?

Subject Procedures:

Subjects will:

* Receive a single treatment session using the VOLNEWMER device.
* Attend follow-up visits over a 12-week period to assess improvements in elasticity and safety.

The primary outcome is the improvement in skin elasticity of the face and cheeks, measured 12 weeks after treatment using the Cutometer R7. Secondary outcomes include the Global Aesthetic Improvement Scale (GAIS). Safety assessments involve monitoring treatment-emergent adverse events (TEAEs) associated with the application of the investigational medical device.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are aged 19 to under 65 at the time of consent.
* Subjects who seek improvement in facial skin elasticity (both cheeks).
* Subjects who agree not to undergo other procedures affecting skin elasticity during the study.
* Subjects who provide written consent and commit to full trial participation.

Exclusion Criteria:

* Subjects with conditions at the investigational device application site (e.g., scars, open wounds, metal stents, or implants, that could affect the trial)
* Subjects with inappropriate skin conditions or treatment history
* Subjects with allergies or predispositions
* Subjects using inappropriate medications that have the potential to increase the risk of bleeding or delay skin healing.
* Subjects with lifestyle or other unsuitable conditions (Smoking history, participation in another interventional clinical trial prior to screening, not agreeing to use medically acceptable contraception, pregnant or breastfeeding women)
* Subjects deemed inappropriate by the investigator

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-11-10 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in Cutometer R7 values | baseline, 12 weeks
  The change in Cutometer R7 values measured on the cheeks at 12 weeks after the application of the investigational medical device compared to baseline will be evaluated.

SECONDARY OUTCOMES:
Change in Cutometer R7 values | baseline, 8 weeks
  The change in Cutometer R7 values measured on the cheeks at 8 weeks after the application of the investigational medical device compared to baseline will be evaluated.
Global Aesthetic Improvement Scale (GAIS) | 4 weeks, 8 weeks, 12 weeks
  The Global Aesthetic Improvement Scale (GAIS) assessed by both the investigator and the subjects at 4, 8, and 12 weeks after the application of the investigational medical device will be evaluated.
  * Minimum and Maximum Values: The GAIS ranges from -1 (worse) to +3 (excellent improvement).
  * Outcome Interpretation: Higher scores indicate a better aesthetic outcome.
Numeric Rating Scale (NRS) for Pain | Baseline, 4 weeks, 8 weeks, 12 weeks
  The subject's pain level at the treatment site will be evaluated using the Numeric Rating Scale (NRS) at the baseline visit and at 4, 8, and 12 weeks after the application of the investigational medical device.
  * Minimum and Maximum Values: The NRS ranges from 0 (no pain) to 10 (worst imaginable pain).
  * Outcome Interpretation: Higher scores indicate worse pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Chung-Ang University Hospital, Dongjak-gu, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No